CLINICAL TRIAL: NCT00747578
Title: Health-Related Quality of Life and Disease-Related Costs: Comparison Between Ankylosing Spondylitis, Rheumatoid Arthritis and Systemic Lupus Erythematosus in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: The Institutional Review Board of Taichung Veterans General Hospital, Taichung Veterans General Hospital
Other Study IDs: C08129
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Ankylosing Spondylitis
Keywords: ankylosing spondylitis (AS), costs,; rheumatoid arthritis (RA),; systemic lupus erythematosus (SLE),; health-related; quality of life (HRQOL); compare; utility; patients
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1: AS patients who fit the modified New York criteria (1984)
  Exclusion criteria :
  1. Patients who have cognitive impairment.
  2. Patients who have overlapping syndrome of any 2 of the 3 rheumatic disease (eg. RA overlapping with SLE).
  3. Patients who are less than 18 years old or older than 65 years old.
  4. Patients who visited rheumatologists in the outpatient clinics of the Division of Rheumatology at Taichung Veterans General Hospital for less than 4 times in 2008.
- 2: RA patients who fit the American College of Rheumatology (ACR) criteria (1987)
  Exclusion criteria :
  1. Patients who have cognitive impairment.
  2. Patients who have overlapping syndrome of any 2 of the 3 rheumatic disease (eg. RA overlapping with SLE).
  3. Patients who are less than 18 years old or older than 65 years old.
  4. Patients who visited rheumatologists in the outpatient clinics of the Division of Rheumatology at Taichung Veterans General Hospital for less than 4 times in 2008.
- 3: SLE patients who fit the ACR revised criteria for the classification of SLE (1997)
  Exclusion criteria :
  1. Patients who have cognitive impairment.
  2. Patients who have overlapping syndrome of any 2 of the 3 rheumatic disease (eg. RA overlapping with SLE).
  3. Patients who are less than 18 years old or older than 65 years old.
  4. Patients who visited rheumatologists in the outpatient clinics of the Division of Rheumatology at Taichung Veterans General Hospital for less than 4 times in 2008.

SUMMARY:
Ankylosing spondylitis (AS), rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE) are the most common rheumatic diseases dealt with rheumatologists in Taiwan. In previous studies, the 3 diseases all have broad impacts on health-related quality of life of patients and drive enormous economic burden on patients and society. The objective of this study is to compare health-related quality of life and disease-related costs between patients with the 3 different diseases.

We will invite at least 100 patients with AS, RA or SLE respectively who are regularly followed in the outpatient clinic of the Division of Rheumatology at Taichung Veterans General Hospital (VGHTC) to participate in the study. Patients who have cognitive impairment, who are older than 65 years old or younger than 18 years old, who have overlapping syndrome of any 2 of the 3 rheumatic diseases (eg. RA overlapping with SLE) or who have visited rheumatologists in the outpatient clinics at VGHTC for less than 4 times in 2008 will be excluded. Patients who agree to take part will attend a comprehensive clinical examination in the outpatient department. Patients will complete a questionaire including demographic and disease characteristics, and health-related quality of life at the time of survey. The questionaires about disease-related costs will be completed once per quarter throughout 2009. The four questionaires about costs will be given at the time of initial survey and will be returned by returned by mail or in the following outpatient clinics visits every 3 months in 2009.

The result of this study will help patients to realize their own health-related quality of life and disease-related costs and help government in Taiwan to realize the socioeconomic burden of the 3 common rheumatic diseases and to allocate health care resources more properly in the future.

ELIGIBILITY:
Inclusion Criteria:

* AS patients who fit the modified New York criteria (1984)
* RA patients who fit the American College of Rheumatology (ACR) criteria (1987)
* SLE patients who fit the ACR revised criteria for the classification of SLE (1997)

Exclusion Criteria:

* 1. Patients who have cognitive impairment.
* 2. Patients who have overlapping syndrome of any 2 of the 3 rheumatic disease (eg. RA overlapping with SLE).
* 3. Patients who are less than 18 years old or older than 65 years old.
* 4. Patients who visited rheumatologists in the outpatient clinics of the Division of Rheumatology at Taichung Veterans General Hospital for less than 4 times in 2008.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will invite at least 100 patients with AS who fit the modified New York criteria (1984) [19] , at least 100 patients with RA who fit the American College of Rheumatology (ACR) criteria (1987) [20] and at least 100 patients with SLE who fit the ACR revised criteria for the classification of SLE (1997) [21] in the outpatient clinics of the Division of Rheumatology at Taichung Veterans General Hospital to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-09

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan